CLINICAL TRIAL: NCT03170310
Title: Apatinib Treatment for Advanced Esophagus Cancer ,One-armed，Exploratory，Openting , Clinical Trail.
Brief Title: Apatinib Treatment for Advanced Esophagus Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HNP006
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Advanced Esophagus Cancer
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib (Experimental)
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib500 mg,po,qd,continuous dosing until PD, death or not tolerated toxicity.

SUMMARY:
Subject ever received a standard chemotherapy solution progression or recurrence or can't tolerate chemotherapy with advanced esophageal squamous carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 to 75 years old, men and women;
* 2. After histopathological and immunohistochemical examination diagnosis of esophageal squamous cell carcinomas. At least one measurable lesion after the treatment (the length to diameter of CT scan≥10 mm , accord with the requirement of RESCIST 1.1);the lesions of whom had not received radiotherapy.
* 3. Advanced esophageal squamous cell carcinoma without molecular targeted drug therapy;
* 4. ECOG PS:0-1;
* 5. Life expectancy≥12 weeks;
* 6. Patients who have disease progressed or relapsed after standard chemotherapy, or who have been unable to tolerate chemotherapy;
* 7. The main organs function properly, that is, meet the following criteria:

  1. blood routine examination: HB≥90 g / L; (without blood transfusion during 14 days) ANC≥1.5×109 /L; PLT≥80×109 / L;
  2. biochemical examination: ALB≥30g / L; (without infusion of albumin during 14 days) ALT and AST<2ULN; TBIL≤1.5ULN; Plasma Cr≤1.5ULN;
* 8. The results of the serum pregnancy test of women in childbearing age must be negative in the 7 days prior to treatment; all patients (both male and female) should take adequate barrier contraception within the entire treatment and 4 weeks after treatment.
* 9. Subject should volunteer to join the study, sign the informed consent, have good compliance and cooperate with the follow-up;
* 10. Investigator believe that subject who can benefit.

Exclusion Criteria:

* 1. In the past or at the same time with suffered from other malignancies;
* 2. Pregnant or lactating women;
* 3. Patients with high blood pressure and can't get a good control after antihypertensive drug therapy (systolic blood pressure>150mmHg, diastolic blood pressure>100mmHg); patients with grade Ⅱ or more myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including QTC interval≥450ms) and Ⅲ~Ⅳ grade cardiac insufficiency according to NYHA; cardiac color Doppler ultrasonography: LVEF <50%;
* 4. Unable to swallow, chronic diarrhea and intestinal obstruction, significantly affect the drug taking and absorption;
* 5. With a clear risk of gastrointestinal bleeding (such as locally active ulcer lesions, fecal occult blood above + +), history of gastrointestinal bleeding within 6 months, and unhealed wounds;
* 6. Central nervous system metastasis has occurred;
* 7. With abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg<2g/L), with bleeding tendency or receiving thrombolytic or anticoagulant therapy;
* 8. With mental illness, or mental history of drug abuse;
* 9. With anastomotic recurrence;
* 10. Patients who have participated in other drug clinical trials in 4 weeks;
* 11. Patients who have concomitant diseases that are seriously compromise the patient's safety or affect the patient to complete the study according to the researcher's judgment;
* 12. Patients those researchers believe not suitable for the inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-02-21 (Estimated); Study Completion 2019-09-21 (Estimated)

PRIMARY OUTCOMES:
Progress free survival | 24 months
  Time subject into the group to tumor objective progression.

SECONDARY OUTCOMES:
Overall survival | up to 24 months
  Time subject into the group to die.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided